CLINICAL TRIAL: NCT03357289
Title: Safety and Efficacy Study of Mix Vaccine in Kidney Cancer Patient
Brief Title: Mix Vaccine for Metastatic Kidney Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Jinan University Guangzhou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: kidney cancer MV
Record Dates: First submitted 2017-11-23; First posted 2017-11-29 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2018-11

CONDITIONS: Metastasis From Malignant Tumor of Kidney (Disorder); Reaction - Mixed Vaccine
MeSH Terms: interventions — Immunotherapy, Active

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mix vaccine (Experimental): In this group, the patients will receive mix vaccine. The check indexes are image examination (CT, MRI or PET scan) and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Biological: Mix vaccine
- Control (No Intervention): In this group, the patients will receive no special treatment and as a control group. The check indexes are image examination (CT, MRI or PET scan) and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).

INTERVENTIONS:
Biological: Mix vaccine — Each treatment: 0.5 ml /week, Subcutaneous injection of the deltoid muscle
  Other Names: Active immunotherapy for cancer
  Arms: Mix vaccine

SUMMARY:
The aim of this study is the safety and efficacy of mix vaccine to small metastases of kidney cancer.

DETAILED DESCRIPTION:
By enrolling patients with small metastases of kidney cancer adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of mix vaccine.

The safety will be evaluated by statistics of adverse reactions. The efficacy will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies after cancer recurrence
* Body tumor 1-6, the maximum tumor length < 2 cm
* KPS ≥ 70, lifespan > 6 months
* Platelet count ≥ 80×109/L，white blood cell count ≥ 3×109/L, neutrophil count ≥ 2×109/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Relief degree of tumors | 3 months
  It will be evaluated by the Response Evaluation Criteria in Solid Tumors（RECIST）

SECONDARY OUTCOMES:
Progress free survival（PFS） | 1 year
  The duration from the beginning of treatment to cancer recurrence or progression
Overall survival（OS） | 3 years
  The duration from the beginning of treatment to patient death

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer institute of Fuda cancer hospital, Guangzhou, Guangdong, China